CLINICAL TRIAL: NCT01569009
Title: Patterns of Physical Activity Levels in Patients With Bronchiectasis: Cross Sectional Study Using Quantitative Methodology
Brief Title: Physical Activity in Bronchiectasis
Acronym: PhAB
Status: Completed | Type: Observational
Sponsor: University of Ulster (Other)
Collaborators: Belfast Health and Social Care Trust (Other); Western Health and Social Care Trust (Other); Southern Health and Social Care Trust (Other Government); Queen's University, Belfast (Other); University of Strathclyde (Other)
Responsible Party: Principal Investigator, Judy Bradley, Reader in Physiotherapy, University of Ulster
Other Study IDs: 11/0085
Record Dates: First submitted 2012-03-16; First posted 2012-04-02 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Physical activity; Activity monitor; Pedometer
MeSH Terms: conditions — Bronchiectasis; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational: Patients are asked to continue with their normal daily activities.

SUMMARY:
The primary aim of this study is to examine the physical activity levels of patients with bronchiectasis.

Subsidiary aims are:

1. To examine whether there is a relationship between the physical activity levels of patients with bronchiectasis and clinical phenotype (disease severity, exercise capacity, quality of life or other symptoms of their disease). The investigators also want to explore the relationship between physical activity levels and readiness to change physical activity behaviour (stages of change, self-efficacy, decisional balance and processes of change).
2. To assess the feasibility and acceptability of the physical activity assessment tools: ActiGraph, ActivPAL, pedometer and the International Physical Activity Questionnaire.

Hypothesis:

Patients with bronchiectasis will have low levels of physical activity, and this is related to their clinical phenotype (disease severity, exercise capacity, quality of life and other symptoms of their disease) and also their readiness to change physical activity behaviour (stages of change, self-efficacy, processes of change and decisional balance).

DETAILED DESCRIPTION:
Bronchiectasis is the presence of abnormal, irreversibly dilated, thick walled bronchi that have not been caused by cystic fibrosis. Promoting physical activity and decreasing inactivity (e.g. sedentary periods of activity such as sitting/lying) has been proposed as a key component of care for chronic disease but there is no research on physical activity in bronchiectasis. There is research describing physical activity in other respiratory populations, however, the disease trajectory and demographic profile of bronchiectasis is sufficiently different to warrant the proposed research specifically in bronchiectasis

The investigators need to explore physical activity in bronchiectasis and also provide specific information on the instruments used to measure physical activity. There are several methods which could be used to assess physical activity including subjective methods (e.g. questionnaires), objective methods (e.g. motion sensors). In this study the investigators are using a range of assessment tools to help determine their usefulness (feasibility and acceptability from the health professional and patient perspective) for quantifying physical activity in bronchiectasis.

This study will also assess patients' readiness to change (stages of change, self efficacy, decisional balance and processes of change). Understanding patients with bronchiectasis readiness to change physical activity behaviour and the links between the other important outcome measures will help to inform a future physical activity intervention specifically in patients with bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years diagnosis of bronchiectasis confirmed by HRCT or CT
* clinically stable (no exacerbation and no significant change in symptoms or medication in the last four weeks)
* sputum bacteriology completed over the past three months

Exclusion Criteria:

* clinically unstable (pulmonary exacerbation or any change in symptoms or medication in the last four weeks)
* current severe haemoptysis
* pregnancy or any other concomitant condition that would prevent participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bronchiecatsis
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Number of steps on the ActiGraph GT3X+ activity monitor | Seven days
  Participants will wear the ActiGraph GT3X+ activity monitor for seven consecutive full days between Visit 1 (Day 0) and Visit 2 (Day 8).

SECONDARY OUTCOMES:
Number of steps on the ActivPAL activity monitor | Seven days
  A sub-group of participants will wear the ActivPAL (n=20). Participants will wear the ActivPAL activity monitor for seven consecutive full days between Visit 1 (Day 0) and Visit 2 (Day 8).
Time spent in physical activity and in sitting using the International Physical Activity Questionnaire | Day 8
  Participants will complete the International Physical Activity Questionnaire at Visit 2 (Day 8). It will be used to measure participants' time spent in physical activity in the last seven days and also to provide self-reported sitting time.
Number of steps on the Yamax Digiwalker pedometer | Seven days
  Participants will wear the Yamax Digiwalker pedometer for seven consecutive full days between Visit 1 (Day 0) and Visit 2 (Day 8).
Exercise Capacity using the Modified Shuttle Test | Day 8
  Participants will complete the Modified Shuttle Test at Visit 2 (Day 8).
Quality of Life using the Quality of Life Questionnaire - Bronchiectasis | Day 8
  Participants will complete the Quality of Life Questionnaire - Bronchiectasis questionnaire at Visit 2 (Day 8).
Quality of Life using the EuroQOL-5D | Day 8
  Participants will complete the EuroQOL-5D at Visit 2 (Day 8).
Quality of Life using the Leicester Cough Questionnaire | Day 8
  Participants will complete the Leicester Cough Questionnaire at Visit 2 (Day 8).
Stage of change in terms of physical activity using the Stages of Change Questionnaire | Day 8
  Participants will complete the Stages of Change Questionnaire at Visit 2 (Day 8). The Stages of Change Questionnaire is the temporal part of the transtheoretical model. It will be used to determine the current stage of change the participant is at in terms of their physical activity behaviour.
Confidence to undertake physical activity using Marcus's Self-Efficacy Questionnaire | Day 8
  Participants will complete Marcus's Self-Efficacy Questionnaire at Visit 2 (Day 8). Marcus's Self-Efficacy Questionnaire is a component of the transtheoretical model which will provide more detailed information on each individual's confidence to undertake physical activity in different situations.
Perception of the benefits and negative aspects of physical activity using Marcus's Decisional Balance Questionnaire | Day 8
  Participants will complete Marcus's Decisional Balance Questionnaire at Visit 2 (Day 8). Marcus's Decisional Balance Questionnaire is a component of the transtheoretical model which will assess each individual's perceptions of the benefits and negative aspects of physical activity.
Strategies used to progress through the different stages of change using Marcus's Processes of Change Questionnaire | Day 8
  Participants will complete Marcus's Processes of Change Questionnaire at Visit 2 (Day 8). Marcus's Processes of Change Questionnaire is a component of the transtheoretical model describing the strategies and techniques individuals use to progress through the different stages of change.
Perception of the feasibility and acceptability of the physical activity outcome measures. | Day 8
  The researcher and the participants will answer the feasibility and acceptability questions at Visit 2 (Day 8). The feasibility and acceptibility questions were designed specifically for this study to assess the researchers' and patients' perspectives of the feasibility and acceptability of the physical activity outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Judy M Bradley, PhD, Principal Investigator — University of Ulster
Locations (3):
- United Kingdom (3):
  - Craigavon Area Hospital, Portadown, Armagh
  - Northern Ireland Regional Respiratory Centre (Belfast City Hospital), Belfast, Co Antrim
  - Altnagelvin Area Hospital, Londonderry, Co Derry

REFERENCES:
- [Derived] O'Neill B, McDonough SM, Wilson JJ, Bradbury I, Hayes K, Kirk A, Kent L, Cosgrove D, Bradley JM, Tully MA. Comparing accelerometer, pedometer and a questionnaire for measuring physical activity in bronchiectasis: a validity and feasibility study? Respir Res. 2017 Jan 14;18(1):16. doi: 10.1186/s12931-016-0497-2. PMID 28088206
- [Derived] Wilson JJ, Kirk A, Hayes K, Bradbury I, McDonough S, Tully MA, O'Neill B, Bradley JM. Applying the Transtheoretical Model to Physical Activity Behavior in Individuals With Non-Cystic Fibrosis Bronchiectasis. Respir Care. 2016 Jan;61(1):68-77. doi: 10.4187/respcare.04154. Epub 2015 Dec 8. PMID 26647454
- [Derived] Bradley JM, Wilson JJ, Hayes K, Kent L, McDonough S, Tully MA, Bradbury I, Kirk A, Cosgrove D, Convery R, Kelly M, Elborn JS, O'Neill B. Sedentary behaviour and physical activity in bronchiectasis: a cross-sectional study. BMC Pulm Med. 2015 May 13;15:61. doi: 10.1186/s12890-015-0046-7. PMID 25967368